CLINICAL TRIAL: NCT06582927
Title: Mindfulness Training for First Responders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Unlikely Collaborators Inc. (Unknown)
Responsible Party: Principal Investigator, Amishi Jha, Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240877
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training Group A (Experimental): Participants in this group will receive mindfulness training in up to 8 weeks.
  Interventions: Behavioral: Mindfulness-Based Attention Training (MBAT)
- Wait-list condition Group B (Active Comparator): Participants in this group will be on a waiting list to receive the identical intervention as the experimental group at a later time. Total participation in the mindfulness training will be 8 weeks
  Interventions: Behavioral: Mindfulness-Based Attention Training (MBAT)

INTERVENTIONS:
Behavioral: Mindfulness-Based Attention Training (MBAT) — MBAT is an evidence-based 8-hour mindfulness program that comprises 4 central topics and associated practices. The concentration topic introduces participants to mindfulness "basics," including discussion of focused attention and mind wandering. The body awareness theme involves the cultivation of greater self-awareness, and the development of equanimity. The open monitoring theme emphasizes awareness of and receptivity to changing experiences and moments of uncertainty. The theme of connection addresses leadership and group cohesion, and the cultivation of kindness and connection with others.
  The course content and materials in the present study will entail the foundational MBAT curriculum and other related content delivered virtually over Zoom but will consist of 8, 1-hour sessions delivered across 8 consecutive weeks.

SUMMARY:
The present study evaluates the efficacy of Mindfulness-Based Attention Training on measures targeting cognitive abilities and emotional well-being in first responders.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 75 years of age
2. Individuals who are fluent English speakers
3. Individuals who are able to adequately and independently use electronic devices, such as a laptop, computer, or tablet, and have Internet connection
4. Individuals who are willing and able to consent to participate in the study
5. Participants in all phases of the study must be individuals who are affiliated with the Los Angeles County Fire Department peer support group.

Exclusion Criteria:

1. Individuals with an active and untreated mental health issue and/or hospitalization for psychological/mental health issues within the past month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in sustained attention | Baseline to week 11
  The Sustained Attention to Response Task (SART) is used to assess attentional performance and mind wandering (i.e., off-task thinking which is typically self-generated and compromises the performance of the task at hand). The task uses a continuous performance paradigm involving button presses to frequently presented nontargets (numbers 0, 1, 2, 4, 5, 6, 7, 8, and 9) but requires the participants to withhold their motor response to the infrequent target (number 3). Withholding responses only to infrequent targets encourages a pre-potent response and mind wandering. Real-time subjective experience of mind wandering during SART is assessed through experience-sampling probes randomly presented throughout the task.
Change in resilience | Baseline to week 11
  Resilience is assessed via the 6-item Brief Resilience Scale (BRS). The scores range from 6 to 30, with a higher score indicating a higher level of resilience.

SECONDARY OUTCOMES:
Change in decentering | Baseline to week 11
  Decentering is assessed via the 11-item decentering sub-scale of the experience questionnaire (EQ-D). The decentering score ranges from 1 to 55, with a higher score indicating a higher level of decentering.
Change in positive affect | Baseline to week 11
  Positive Affect is assessed with the 5-item positive sub-scale from Positive and Negative Affect Schedule (PANAS). PANAS Positive has a range of scores from 5 to 25, with a higher score indicating a higher positive mood.
Change in negative affect | Baseline to week 11
  Negative Affect is assessed with the 5-item negative sub-scale from Positive and Negative Affect Schedule (PANAS-10). PANAS Negative has a range of scores from 5 to 25, with a higher score indicating a higher negative mood.
Change in perceived stress | Baseline to week 11
  Perceived stress is assessed with the 4-item Perceived Stress Scale (PSS-4). PSS-4 has a range of scores from 0 to 16, with a higher score indicating a higher level of perceived stress.
Change in burnout | Baseline to week 11
  Burnout is assessed with the 12-item Burnout Assessment Tool (BAT-12). BAT-12 has a range of score from 1 to 5, with a higher score indicated a higher level of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No